CLINICAL TRIAL: NCT00288847
Title: Functional Surface Electromyogram of Knee Extensors in Healthy Humans and Patients With Patella-dislocation.
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Lab. for Orthopaedic Biomechanics, University of Basel (Other); University Children's Hospital Basel (Other)
Responsible Party: Sponsor
Other Study IDs: LOB_00001_patella
Record Dates: First submitted 2006-02-02; First posted 2006-02-08 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Patella-Dislocation
Keywords: Patella Dislocation; Surface EMG; Gender difference
MeSH Terms: conditions — Patellar Dislocation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The activation of the knee extensors in adults after patella dislocation.

The kneecap can dislocate due to an accident or also only due to an interior turn in the stretched knee joint out of its sliding bearing. E. Arendt (Arendt 2002) wrote an overview work, in which possible causes and working methods to the patella dislocation are discussed. Despite almost one hundred quotations the authors are not able find the causes and the possible treatment concepts. The study will examined healthy adults (25 female and 25 men) and 25 patients with patella dislocation by a routine applied clinical gait analysis and surface EMG (after the European SENIAM guidelines) iin the Laboratory for Gait Analysis Basel of the Children's University Hospital Basel. The combination of gait analysis and the surface EMG with Wavelet analysis may objectify possible reasons for a patella dislocation

DETAILED DESCRIPTION:
Introduction The kneecap can dislocate due to an accident or also only due to an interior turn in the stretched knee joint out of its sliding bearing. E. Arendt (Arendt 2002) wrote an overview work, in which possible causes and working methods to the patella dislocation are discussed. Despite almost one hundred quotations the authors are not able find the causes and the possible treatment concepts. The study will examined healthy adults (25 female and 25 men) and 25 patients with patella dislocation by a routine applied clinical gait analysis and surface EMG (after the European SENIAM guidelines) in the Laboratory for Gait Analysis Basel of the Children's University Hospital Basel. The combination of gait analysis and the surface EMG with Wavelet analysis may objectify possible reasons for a patella dislocation and compare the intensity pattern of the EMG between the groups.

Method All subjects (healthy and patients with a patella dislocation) will be prior to the study informed about the study and sign the consent from

The investigation will include the following tasks:

* Preparation of the subject for a clinical gait analysis with placing reflecting marker on the lower body according to the maker setup of Davis et al. (Davis III et al., 1991.
* Preparation of the subject for a surface EMG of the muscles: gastrocnemius medialis, tibialis anterior, vastus medialis, vastus lateralis, rectus femoris, biceps femoris, semitendinosus according to the SENIAM-Standard.
* Measurements: 10 trials of level walking in self selected speed and 3 times 5 single leg quads on the force plate.
* System: VICON 460 (6 Cameras, 120 Hz, Oxford Metrics Ltd., UK).
* EMG-System: Zebris, Tuebingen, Germany; Amplifiers: Biovision, Wehrheim, Germany, EMG-Electrodes: Bipolar Ag/AgCl Surface Electrodes Noraxon, Sampling rate: 2520 Hz
* Data analysis: Kinetic-and kinematic data with the Vicon-Software, EMG-Data with Wavelet Package (Biomechanigg, Calgary, Canada)
* Statistical Analysis: ANVOA

ELIGIBILITY:
Inclusion Criteria:

* Patient: Patella Dislocation before surgery
* Control: healthy

Exclusion Criteria:

* Patient: Patella Dislocation not able to walk,
* Patient: using orthosis or crutches
* Control: knee injury (e.g. ACL-rupture)
* Control: leg surgery in the last 5 years
* Control: sport injury in the last 6 month (e.g. Muscle pulling)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Goepfert, MEng, Principal Investigator — Lab. for Orthopaedic Biomechanics, University of Basel; Dieter Wirz, MD, Principal Investigator — Lab. for Orthopaedic Biomechanics, University of Basel; Alma U Daniels, Ph.D., Study Chair — Lab. for Orthopaedic Biomechanics, University of Basel
Locations (1):
- Lab. for Orthopaedic Biomechanics, University of Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Background] Von Tscharner V, Goepfert B. Estimation of the interplay between groups of fast and slow muscle fibers of the tibialis anterior and gastrocnemius muscle while running. J Electromyogr Kinesiol. 2006 Apr;16(2):188-97. doi: 10.1016/j.jelekin.2005.07.004. Epub 2005 Sep 1. PMID 16139523
- [Background] von Tscharner V, Goepfert B. Gender dependent EMGs of runners resolved by time/frequency and principal pattern analysis. J Electromyogr Kinesiol. 2003 Jun;13(3):253-72. doi: 10.1016/s1050-6411(02)00111-6. PMID 12706605
- [Background] von Tscharner V, Goepfert B, Nigg BM. Changes in EMG signals for the muscle tibialis anterior while running barefoot or with shoes resolved by non-linearly scaled wavelets. J Biomech. 2003 Aug;36(8):1169-76. doi: 10.1016/s0021-9290(03)00086-1. PMID 12831743
- [Background] von Tscharner V, Gopfert B, Wirz D, Friederich NF. [Analysis of wavelet transformed electromyographic signals that were altered by wearing a knee brace]. Biomed Tech (Berl). 2004 Mar;49(3):43-8. doi: 10.1515/BMT.2004.009. German. PMID 15106897
- [Background] von Tscharner V. Time-frequency and principal-component methods for the analysis of EMGs recorded during a mildly fatiguing exercise on a cycle ergometer. J Electromyogr Kinesiol. 2002 Dec;12(6):479-92. doi: 10.1016/s1050-6411(02)00005-6. PMID 12435545
- [Background] von Tscharner V. Intensity analysis in time-frequency space of surface myoelectric signals by wavelets of specified resolution. J Electromyogr Kinesiol. 2000 Dec;10(6):433-45. doi: 10.1016/s1050-6411(00)00030-4. PMID 11102846